CLINICAL TRIAL: NCT05656586
Title: Mechanisms and Effects of Pallidal Deep Brain Stimulation on Levodopa Resistant Motor Signs in Parkinson's Disease; Udall Project 2 Aim 2A&C
Brief Title: Udall Project 2 Aim 2A&C
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00016988
Record Dates: First submitted 2022-12-05; First posted 2022-12-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Participants: Inclusion criteria for all aims/experiments
  * Receiving DBS therapy in GP or STN for treatment of PD
  * Implanted with Medtronic Percept DBS system
  * At least 3 months since initial activation of the neurostimulator
  Interventions: Other: observational-- no intervention

INTERVENTIONS:
Other: observational-- no intervention — observational

SUMMARY:
This protocol will leverage the novel (on-label, FDA-approved) local field potential measuring capability of the Medtronic Percept™ PC or RC DBS system to study the effects of globus pallidus internus, globus pallidus externus (GPi, GPe), and subthalamic nucleus (STN) DBS on: the wash-out and wash-in dynamics of motor behavior and local field potentials (LFPs) and correlations between fluctuations in gait and LFPs during activities of daily living (recorded over a minimum of 4 weeks). These experiments will elucidate the relationships between LFPs oscillations, lower limb function, postural control and gait performance.

DETAILED DESCRIPTION:
This protocol will leverage the novel (on-label, FDA-approved) local field potential measuring capability of the Medtronic Percept™ PC or RC DBS system to study the effects of globus pallidus internus, globus pallidus externus (GPi, GPe), and subthalamic nucleus (STN) DBS on: the wash-out and wash-in dynamics of motor behavior and local field potentials (LFPs) and correlations between fluctuations in gait and LFPs during activities of daily living (recorded over a minimum of 4 weeks). These experiments will elucidate the relationships between LFPs oscillations, lower limb function, postural control and gait performance.

ELIGIBILITY:
Inclusion Criteria:

* Receiving DBS therapy in GP for treatment of PD
* Implanted with Medtronic Percept DBS system
* At least 3 months since initial activation of the neurostimulator
* For the "At Home" experiment only: participants with DBS settings that are sensing compatible.

Exclusion Criteria:

* history of musculoskeletal disorders that significantly affects the ability to perform the motor tasks in the specific experiment in question
* history of dementia or cognitive impairment
* other significant neurological disorder as determined by the PI
* post-operative complications or adverse effects (e.g. ON stimulation dystonias) that affect patient safety or confound the experiment
* lack of capacity to consent (as identified by MaCAT-CR)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Receiving DBS therapy in GP for treatment of PD
  * Implanted with Medtronic Percept DBS system
  * At least 3 months since initial activation of the neurostimulator
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Peak negative power | 30 day
  A servo-controlled ankle manipulandum will be used to obtain objective measures of resistance about the dorsiflexion/plantar flexion axis (range of motion approximately 5 deg. dorsiflexion to 30 deg. plantar flexion; frequency = 1.5 Hz). Two conditions will be tested: passive movement with and without an activation maneuver on the contralateral side (repetitive tapping of the toe or heel).
Stride length | 30 days
  The spatial and temporal parameters of overground steady-state gait will be assessed in the lab or derived from the wearable device (mPower)
Alpha power during standardized daily gait assessment | 30 days
  The participant will use their DBS device patient programmer to record a time stamp and capture LFPs using the implanted Medtronic Percept™ device during the standardized daily gait assessments.
cadence | 30 days
  The spatial and temporal parameters of overground steady-state gait will be assessed in the lab or derived from the wearable device (mPower)

SECONDARY OUTCOMES:
gait speed | 30 days
  The spatial and temporal parameters of steady-state gait will be assessed using a computerized walkway.
time spent away from home | 30 days
  time spent away from home, as measured by the mPower smartphone app
distance traveled from home | 30 days
  distance traveled away from home, as measured by the mPower smartphone app
alpha power immediately following freezing of gait episodes, falls and other major events | 30 days
  The participant will use their DBS device patent programmer to record a time stamp when they experience a freezing of gait episode and LFPs will be recorded immediately following that time by the implanted Medtronic Percept™ device
Peak power of local field potential oscillations | 30 days
  average daytime peak alpha and beta power derived from power spectral density analysis of the local field potential signal recorded by the implanted Medtronic Percept™ device
stride time variability | 30 days
  The spatial and temporal parameters of steady-state gait will be assessed using a computerized walkway.
step length variability | 30 days
  The spatial and temporal parameters of steady-state gait will be assessed using a computerized walkway.

OTHER OUTCOMES:
gait asymmetry | 30 days
  The spatial and temporal parameters of steady-state gait will be assessed using a computerized walkway.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States